CLINICAL TRIAL: NCT01487421
Title: The Physiological Therapy of Type 2 Diabetes - NovoRapid® FlexPen® Before Meals, Additionally Levemir® FlexPen® in the Evening or at Bedtime if Needed
Brief Title: An Observational Study of Insulin Aspart and, if Necessary, Insulin Levemir (FlexPen®) in the Evening or at Bedtime
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: ANA-1934
Record Dates: First submitted 2011-11-25; First posted 2011-12-07 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart; Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SIT
  Interventions: Drug: insulin aspart; Drug: insulin detemir

INTERVENTIONS:
Drug: insulin aspart — Subjects were observed over a time period of 12 weeks after initiation of a supplementary insulin therapy regimen (SIT) with insulin aspart at mealtimes. Administrated subcutaneously (s.c., under the skin)
Drug: insulin detemir — Insulin detemir were added to insulin aspart in the evening or at bedtime, if needed. Administrated subcutaneously (s.c., under the skin)

SUMMARY:
This study is conducted in Europe. The aim of this study is investigate the potential of a supplementary insulin therapy regimen (SIT) as intensification for insufficiently controlled patients with type 2 diabetes in a normal diabetes care setting.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* OAD monotherapy
* OAD combination therapy
* Therapy with OAD and basal insulin
* Conventional insulin therapy with premixed insulin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with insufficiently controlled type 2 diabetes mellitus treated with diet, OAD (oral anti-diabetes drug), long acting insulin, premixed insulin or a combination
Sampling Method: Non-Probability Sample
Enrollment: 2134 (Actual)
Dates: Start 2003-07; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycosylated haemoglobin)

SECONDARY OUTCOMES:
Fasting blood glucose (FBG)
2-hours postprandial blood glucose
Hypoglycemia
Weight development
Adverse Drug Reactions (ADRs) including Serious Adverse Drug Reactions (SADRs)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Mainz, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com